CLINICAL TRIAL: NCT06658496
Title: Development of a Novel Kidney-focused Approach to Treatment of a Patent Ductus Arteriosus (PDA) in Vulnerable Preterm Neonates - A Pilot Study
Brief Title: PDA for Kidneys Study
Acronym: PDA4K
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-1052; A536757 (Other: UW- Madison); Protocol Version 2/10/25 (Other: UW- Madison)
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-05

CONDITIONS: Patent Ductus Arteriosus; Congenital Heart Disease
Keywords: neonate
MeSH Terms: conditions — Ductus Arteriosus, Patent; Heart Defects, Congenital | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neonates with PDA
  Interventions: Device: Near Infrared Spectroscopy

INTERVENTIONS:
Device: Near Infrared Spectroscopy — Application of regional NIRS sensors to brain and kidney sites in the first 72 hours after birth to monitor regional tissue oxygenation.
  Other Names: NIRS

SUMMARY:
The goal of this observational study is to gather more information on kidney oxygen levels in babies with a patent ductus arteriosus (PDA), and evaluate the relationships between kidney oxygen levels, PDA status and kidney injury.

Researchers will do this by looking at ultrasound images of the heart, analyzing substances in the urine, and evaluating oxygen levels in the kidneys.

ELIGIBILITY:
Inclusion Criteria:

* Delivered at <32 weeks' gestation
* ≤72 hours of age
* Inpatient at Meriter Hospital, Inc. NICU
* At least one parent/guardian is able to provide parental permission in English or Spanish

Exclusion Criteria:

* Major congenital anomalies of kidney
* Attending physician's discretion to not place NIRS sensors due to clinical concerns
* In the PI or Co-I's medical opinion, there is a significant likelihood that the neonate would not survive the first 3 days of life
* Birth parent aged <18

Ages: 1 Minute to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates born <32 weeks gestational age (GA) at Meriter Hospital, Inc. and outborn neonates admitted to Meriter Hospital, Inc. within 12 hours of life.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Comparison of patent ductus arteriosus (PDA) echocardiography parameters to kidney hypoxia | Days 1 to 7 of age
  Measured through continuous renal near infrared spectroscopy (NIRS) monitoring in neonates with a PDA to those without. Echos will be obtained every 48 hours during the first 7 days of age for a maximum of 3. RSO2 will be recorded until 7 days of age.

SECONDARY OUTCOMES:
Correlation of Iowa PDA score to kidney hypoxia | Days 1-7 of age
  The Iowa PDA score will be classified as low (0-3), moderate (4-6), or high volume (>6) for each echo obtained. Lower scores are optimal. RSO2 correlation will be made with PDA score during the first 7 days of age.
Correlation between urinary biomarkers and Iowa PDA score | Days 1-7 of life
  The Iowa PDA score will be classified as low (0-3), moderate (4-6), or high volume (>6). Urinary NGAL, cystatin C, and beta 2 micro globulin levels will be measured daily for the first 7 days of age and a correlation with the Iowa PDA score to levels of these biomarkers will be made.
Correlation between rates of hypertension and Iowa PDA score | Duration of hospitalization, up to 6 months
  The Iowa PDA score will be classified as low (0-3), moderate (4-6), or high volume (>6). Hypertension will be assessed for throughout hospitalization and a correlation with Iowa PDA score and the diagnosis of hypertension will be made.
Correlation between rates of acute kidney injury (AKI) and Iowa PDA score | Duration of hospitalization, up to 6 months
  The Iowa PDA score will be classified as low (0-3), moderate (4-6), or high volume (>6). The diagnosis of AKI will be made using either or both urine output criteria or serum creatinine criteria and a correlation will be made with the IOWA PDA score in the first 7 days of age.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Harer, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Meriter Hospital, Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No